CLINICAL TRIAL: NCT06791759
Title: The Effects of the Course on Technology Use in Nursing on Students' Self-directed Learning Readiness and Attitudes Toward Technology: A Quasi-experimental Study
Brief Title: The Effects of the Course on Technology Use in Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma DURSUN ERGEZEN, Assistant Professor, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FatmaErgezen
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Nursing Student; Technology; Self Directed Learning
MeSH Terms: interventions — Nursing

STUDY DESIGN:
Intervention Model Description: This was a quasi-experimental study employing a pretest-posttest design with a control group. The participants consisted of first-year nursing students enrolled in the spring semester of the 2023-2024 academic year at a nursing faculty in Türkiye. Students who attended the course on the technology use in nursing were included in the intervention group. The course on the technology use in nursing is an elective course. It consisted of 2 hours per week over 14 weeks. Students in the control group attended the 'Health Assessment' course, which is based on the Functional Health Patterns Model.
Masking Description: The statistician was masked in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The course on technology use in nursing (Experimental): Students attended in the course technology use in nursing. The course consisted of 2 hours per week over 14 weeks. The course aims to provide students with an understanding of fundamental technological developments in nursing, highlighting the importance and impact of technology in nursing education and practice.Theoretical lessons were delivered by two nurse educators over 8 weeks through PowerPoint presentations and interactive discussions. For the remaining five weeks, students were given some assignments to increase their interaction with digital technological tools. Three assignments were planned for each of the students. In this context, microsoft teams, canva, microsoft powerpoint, kahoot, mentimeter, quizlet, ed-puzzle, capcut, mobile health applications, google classroom, discord and artificial intelligence applications were used for assignments.
  Interventions: Other: The course on technology use in nursing
- Control (No Intervention): Students in the control group attended the 'Health Assessment' course, which is based on the Functional Health Patterns Model. Various assignments were given to students within the scope of this course. Students were divided into groups, prepared patient interview questions for each pattern, and conducted role-play interviews. Students did not use any digital tools within the scope of the course assignments.

INTERVENTIONS:
Other: The course on technology use in nursing — Students attended in the course technology use in nursing. The course consisted of 2 hours per week over 14 weeks. The course aims to provide students with an understanding of fundamental technological developments in nursing, highlighting the importance and impact of technology in nursing education and practice.Theoretical lessons were delivered by two nurse educators over 8 weeks through PowerPoint presentations and interactive discussions. For the remaining five weeks, students were given some assignments to increase their interaction with digital technological tools. Three assignments were planned for each of the students. In this context, microsoft teams, canva, microsoft powerpoint, kahoot, mentimeter, quizlet, ed-puzzle, capcut, mobile health applications, google classroom, discord and artificial intelligence applications were used for assignments.
  Arms: The course on technology use in nursing

SUMMARY:
This study aimed to examine the effect of the course on technology use in nursing on students' readiness for self-directed learning (SDLR) and attitudes toward technology. Research hypotheses are as follows:

* H1-1: The course on technology use in nursing affects nursing students' SDLR.
* H1-2: The course on technology use in nursing affects nursing students' attitudes toward technology.

DETAILED DESCRIPTION:
The study has a quasi-experimental design. In the study, the intervention group participated in a 14-week course titled "Technology Use in Nursing," consisting of 2-hour weekly sessions. On the other hand, the control group attended a 14-week course titled "Health Assessment," also consisting of 2-hour sessions per week. Participants in the intervention group were given various tasks to enhance integration with technology. Students used various digital tools (such as Edpuzzle, artificial intelligence programs, mobile health applications, etc.). In the control group, participants were assigned the task of conducting interviews based on the Functional Health Patterns model in group work settings. No tasks involving digital tools were assigned to students in the control group.

Students were invited to participate in the study, and assignments to groups were made. After the group assignments, pre-tests were administered using the "Self-Directed Learning Readiness Scale" and the "Attitudes Toward Technology Survey." Post-tests were collected using the same scales at the end of the courses (week 14).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Enrollment in one of the elective courses: 'Technology use in nursing' or 'health assessment'
* Taking elective courses for the first time

Exclusion Criteria:

* Refusal to participate in the study at any stage of the research process
* Incomplete completion of the data collection forms

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Self-directed Learning Readiness | Data were collected at two different time points in the study: first after students agreed to participate in the study (week 2 of the course), and second at the end of the course (week 14).
  The self-directed learning readiness was measured with Self-Directed Learning Readiness Scale (SDLR) . The SDLRS consists of 40 items and uses a five-point Likert scale. The scale includes three sub-dimensions: self-management, willingness to learn, and self-control. The total score ranges from a minimum of 40 to 200 points. A total score 150 is recommended as the cut-off point for determining SDLR. As the total score increases, it is assumed that the student's SDL ability also increases.
Attitudes toward technology | Data were collected at two different time points in the study: first after students agreed to participate in the study (week 2 of the course), and second at the end of the course (week 14).
  The technology attitudes of students was measured with Technology Attitude Scale. The scale consists of 15 items and uses a 6-point Likert scale. The scale includes two sub-dimensions: confidence in and the benefits of using technology and lack of self-efficacy in the use of technology. The total score ranges from a minimum of 15 to a maximum of 90 points. As the total score increases, it is assumed that the student's positive attitudes toward technology also increases.

CONTACTS AND LOCATIONS:
Overall Officials: FATMA Dursun Ergezen, PhD, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol